CLINICAL TRIAL: NCT06236490
Title: Validation of Blood Oxygen Level Test in Well-trained Athletes
Status: Completed | Type: Observational
Sponsor: Institute of Sport - National Research Institute, Poland (Other)
Responsible Party: Principal Investigator, Tomasz Kowalski, Principal Investigator, Institute of Sport - National Research Institute, Poland
Other Study IDs: InstSportPoland
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Athletic Performance
Keywords: bolt; blood oxygen level test; chemosensitivity; baroreceptor sensitivity
MeSH Terms: interventions — Exercise Test

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Particpants - Speedskating Athletes: All the study participants were members of the Polish National Development Team or Polish National Elite Team in either long-track or short-track speedskating. Inclusion criteria were as follows: a valid medical certificate for competitive speedskating, a minimum of six years of training, and no prior exposure to respiratory or respiratory muscle training. Exclusion criteria were as follows: any chronic medical conditions, recent acute medical conditions within the last 4 weeks, COVID-19 infection within the last 6 months, recent stay in an altitude over 1500 meters above sea level within the last 4 weeks, and the use of any ongoing medications.
  Interventions: Diagnostic Test: Blood Oxygen Level Test; Diagnostic Test: Wingate Anaerobic Test; Diagnostic Test: Cardiopulmonary Exercise Test

INTERVENTIONS:
Diagnostic Test: Blood Oxygen Level Test — The study participants rested for 15 minutes before measuring the BOLT score. During this time they were carefully instructed on how to perform the measurement. It was underlined that we do not measure how long one can hold their breath, but the time it takes for the body to react to lack of air and feel the desire to breathe. After a few normal breaths through the nose, after the exhalation, the participants held their breath until they felt the first definite desire to breathe or felt the first involuntary contractions of the respiratory muscles. The first was assessed by the participants, the latter was also visually assessed by the researchers. The nose was closed with the fingers to prevent any gas exchange. The researchers measured the time with a Finis 3x300M stopwatch (FINIS USA, Livermore, CA, USA). Time in seconds, to one decimal place, was noted as a BOLT score. The visualisation of BOLT is presented in Figure 2.
Diagnostic Test: Wingate Anaerobic Test — WAnT was conducted with Monark 874E Cycle Ergometer (Monark Exercise AB, Sweden). Before WAnT, the participants performed a 5-minute warm-up with resistance ranging from 0.8 to 1.2 W/kg. Next, the participants performed a maximal 6-second sprint, with the resistance adjusted to 7.5% of the individual body mass. After a rest interval of 2 to 5 minutes, the participants underwent a 30-second WAnT with resistance set at 7.5% of the individual body mass. They were instructed to attain the highest peak power output as quickly as possible and maintain the highest power output throughout the entire duration of the test. The participants received motivating and enthusiastic verbal support. The following indices were measured and included in the further analysis: peak power (Ppeak), total work (TW), WSSR. All the indices were calculated with the dedicated software (MCE 6.0, JBA Z. Staniak, Poland) linked to the cycle ergometer.
Diagnostic Test: Cardiopulmonary Exercise Test — CPET was performed with the Cortex Metamax B3 (Cortex Biophysik GmbH, Leipzig, Germany), breath-by-breath method, and Cyclus II Ergometer (RBM, Leipzig, Germany). Participants underwent an incremental ramp test, commencing at 55-70W and incrementally increasing the load by 0.17-0.28 W·sec-1, individually adjusted for body mass. The participants were instructed to continue the effort until total exhaustion. All the participants fulfilled the maximum effort criteria (Wiecha et al. 2023): 1) respiratory exchange ratio ≥ 1.10, (2) present VO2 plateau (growth < 100 mL·min-1 in VO2 despite increased cycling power), (3) respiratory frequency ≥ 45 breaths·min-1, (4) declared subjective exertion intensity during CPET ≥ 18 according to the Borg Scale (Borg 1998), (5) blood lactate concentration ≥8 mmol·L-1, (6) peak heart rate ≥ 15 beats·min-1 below predicted maximal heart rate (HRmax) (Lach et al. 2021).

SUMMARY:
Blood Oxygen Level Test (BOLT) was never scientifically validated. Therefore, we investigated the association of BOLT scores with athletic performance in well-trained athletes. The study focuses on exercise tolerance in severe and extreme intensity domains, as they provoke significant homeostatic perturbations.

We perform Wingate Anaerobic Test and Cardiopulmonary Exercise Test, which are part of the regular National Team athletes screening in our lab, to see if the results may be assocciated with BOLT results.

The performance tests are used by the Speedskating National Team multiple times per year as training monitoring and performance assessments of the athletes.

DETAILED DESCRIPTION:
The investigated group consisted of 49 well-trained speedskaters recruited with convenience sampling (out of 58 that volunteered to participate in the study). All the study participants were members of the Polish National Development Team or Polish National Elite Team in either long-track or short-track speedskating. Inclusion criteria were as follows: a valid medical certificate for competitive speedskating, a minimum of six years of training, and no prior exposure to respiratory or respiratory muscle training. Exclusion criteria were as follows: any chronic medical conditions, recent acute medical conditions within the last 4 weeks, COVID-19 infection within the last 6 months, recent stay in an altitude over 1500 meters above sea level within the last 4 weeks, and the use of any ongoing medications. The required sample size was calculated with G* Power (version 3.1.9.2; Germany), with effect size ƒ² = 0.35, level of significance set at α = 0.05, power (1 - β) = 0.95, and number of predictors = 1 (Linear multiple regression: Fixed model, R² deviation from zero). According to the calculations, the required total sample size was 40 participants. In our study, 58 participants were recruited to account for possible dropouts. Finally, 49 participants completed all the required procedures and were included in further analysis.

Three tests are used in the study:

Blood Oxygen Level Test (BOLT) was performed according to The Oxygen Advantage guidelines. The study participants rested for 15 minutes before measuring the BOLT score. During this time they were carefully instructed on how to perform the measurement. It was underlined that we do not measure how long one can hold their breath, but the time it takes for the body to react to lack of air and feel the desire to breathe. After a few normal breaths through the nose, after the exhalation, the participants held their breath until they felt the first definite desire to breathe or felt the first involuntary contractions of the respiratory muscles. The first was assessed by the participants, the latter was also visually assessed by the researchers. The nose was closed with the fingers to prevent any gas exchange. The researchers measured the time with a Finis 3x300M stopwatch (FINIS USA, Livermore, CA, USA). Time in seconds, to one decimal place, was noted as a BOLT score.

Wingate Anaerobic Test (WAnT) was conducted with Monark 874E Cycle Ergometer (Monark Exercise AB, Sweden). Before WAnT, the participants performed a 5-minute warm-up with resistance ranging from 0.8 to 1.2 W/kg. Next, the participants performed a maximal 6-second sprint, with the resistance adjusted to 7.5% of the individual body mass. After a rest interval of 2 to 5 minutes, the participants underwent a 30-second WAnT with resistance set at 7.5% of the individual body mass. They were instructed to attain the highest peak power output as quickly as possible and maintain the highest power output throughout the entire duration of the test. The participants received motivating and enthusiastic verbal support. The following indices were measured and included in the further analysis: peak power (Ppeak), total work (TW), WSSR. All the indices were calculated with the dedicated software (MCE 6.0, JBA Z. Staniak, Poland) linked to the cycle ergometer.

Cardiopulmonary Exercise Testing (CPET) was performed with the Cortex Metamax B3 (Cortex Biophysik GmbH, Leipzig, Germany), breath-by-breath method, and Cyclus II Ergometer (RBM, Leipzig, Germany). Participants underwent an incremental ramp test, commencing at 55-70W and incrementally increasing the load by 0.17-0.28 W·sec-1, individually adjusted for body mass. The participants were instructed to continue the effort until total exhaustion. All the participants fulfilled at least five out of the six maximum effort criteria as follows: 1) respiratory exchange ratio ≥ 1.10, (2) present VO2 plateau (growth < 100 mL·min-1 in VO2 despite increased cycling power), (3) respiratory frequency ≥ 45 breaths·min-1, (4) declared subjective exertion intensity during CPET ≥ 18 according to the Borg Scale, (5) blood lactate concentration ≥8 mmol·L-1, (6) peak heart rate ≥ 15 beats·min-1 below predicted maximal heart rate (HRmax) . The following indices were measured with 15 second intervals and included in the further analysis: maximum oxygen uptake (VO2max) in mL·min-¹·kg-¹, and time from achieving VO2max to the cessation of the test (TtC) in seconds.

All the athletes were familiarised with testing procedures, as they peformed them multiple times before. The medical screening is performed on a testing day in the morning. All the athletes have to undergone the medical screening.

Further, the performance test results will be used to validate BOLT test in terms of association with athletic performance.

ELIGIBILITY:
Inclusion criteria were as follows:

* a valid medical certificate for competitive speedskating,
* a minimum of four years of competitive training,
* no prior exposure to respiratory or respiratory muscle training.

Exclusion criteria were as follows:

* any chronic or acute medical condition within the last 4 weeks,
* recent stay at an altitude over 1500 meters above sea level within the last 4 weeks,
* the use of any ongoing medications, smoking, any ongoing allergy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Elite Speedskaters, Members of the National Team
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Blood Oygen Level Score | June-September 2023
  Voluntary breatholding untill the first signs of discomfort of respiratory muscle contraction, measured in seconds.
Wingate Test Result - total completed work | June-September 2023
  Total work completed during Wingate 30 second test, measured in kilojouls
Maximal Oxygen Uptake - VO2max | June-September 2023
  Maximal oxygen uptake, measured in ml/kg/min.
Time to cessation during cardiopulmonary testing | June-September 2023
  Time in seconds from achieving oxygen uptate plateau to cessation of exercise.
Wingate Test Result - peak power | June-September 2023
  Peak power during Wingate 30 second test, measured in watts.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Sport - National Research Institute, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No